CLINICAL TRIAL: NCT01094119
Title: A Randomized Comparison of Intraoperative Warming With the LMA PerfecTemp and Forced-air
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-146
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Warming Systems During Surgery
Keywords: heated blanket; heated pad

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bair Hugger heated blanket (Active Comparator): Patients will be warmed during surgery with the Bair Hugger heated blanket.
  Interventions: Device: heated blanket
- LMA PerfecTemp system (Active Comparator): Patients will be warmed during surgery with the PerfecTemp heated pad .
  Interventions: Device: heated pad

INTERVENTIONS:
Device: heated blanket — heated blanket
  Other Names: Bair Hugger
  Arms: Bair Hugger heated blanket
Device: heated pad — patients will be warmed with a heated pad during surgery.
  Other Names: LMA PerfecTemp system
  Arms: LMA PerfecTemp system

SUMMARY:
Recently, a novel posterior heating system has been developed that provides enhanced pressure relief: the Laryngeal Mask Airway (LMA) PerfecTemp. Anactodal experience with this FDA-approved system suggests that the PerfecTemp warmer is effective, even in open abdominal surgery. The investigators therefore propose to test the hypothesis that intraoperative distal esophageal (core) temperatures with PerfecTemp warming are non-inferior to upper-body forced-air warming in patients undergoing open major abdominal surgery under general anesthesia.

Secondary hypotheses include that:

1. intraoperative core temperatures are superior with PerfecTemp than upper-body forced-air warming
2. final intraoperative core temperature is non-inferior with PerfecTemp than upper-body forced-air warming
3. final intraoperative core temperature is superior with PerfecTemp than upper-body forced-air warming.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index 20-36 kg/m2
* Age 18-75 yrs
* ASA Physical Status 1-3
* Supine position (with or without lithotomy)

Exclusion Criteria:

* Pre-operative fever
* Serious skin lesions
* And contraindication to either PerfecTemp or forced-air warming

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bair Hugger Heated Blanket | LMA PerfecTemp System
Started | 34 | 36
Completed | 32 | 32
Not Completed | 2 | 4
Not completed — Lack of Efficacy | 2 | 4

BASELINE CHARACTERISTICS:
Population: Most baseline characteristics were well balanced be- tween the randomized groups. However, patients assigned to resistive heating were more likely to have higher ASA physical status classification. Thus, ASA status was adjusted for in all analyses. Patients in each warming group were given comparable doses of volatile anesthesia and opioid.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bair Hugger Heated Blanket | LMA PerfecTemp System | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 51 (15) | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 15 | 12 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 34 | 34 | 68
  Not Caucasian | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46
  Canada | 11 | 13 | 24
preoperative oral temperature [Mean (Standard Deviation); unit: degrees C] | 36.2 (.9) | 36.8 (.8) | 36.2 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average Core Temperature
Description: Time weighted average core temperature (esophogeal temperature) from tracheal intubation to 3 hours after or tracheal extubation
Time Frame: from tracheal intubation to 3 hours after or tracheal extubation
Population: Randomized patients.
Measure: Mean (Standard Deviation); unit: Degrees C
Arm/Group | Bair Hugger Heated Blanket | LMA PerfecTemp System
Number analyzed (Participants) | 34 | 36
Degrees C | 36.11 (.5) | 36.02 (.55)

2. Secondary Outcome: Proportion of Patients With Temperatures Above 36 Degree
Description: Proportion of patients with esophogeal temperatures above 36 degree at the end of surgery
Time Frame: at the end of surgery
Population: Enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Bair Hugger Heated Blanket | LMA PerfecTemp System
Number analyzed (Participants) | 34 | 36
Participants | 30 | 21
Statistical Analysis 1: Comparison: Bair Hugger Heated Blanket vs LMA PerfecTemp System; Test type: Superiority; p = 0.0069, Regression, Logistic

ADVERSE EVENTS:
Time Frame: In-hospital
Arm/Group | Bair Hugger Heated Blanket | LMA PerfecTemp System
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 0/34 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No